CLINICAL TRIAL: NCT06641635
Title: A Multicenter, Non-inferiority, Phase 3, Randomized Controlled Study of Moderated Hypofractionated Online Adaptive Radiotherapy for Cervical Cancer
Brief Title: Moderated Hypofractionated Online Adaptive Radiotherapy in Cervical Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Shandong Cancer Hospital and Institute (Other); Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWIFT-1
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-10

CONDITIONS: Cervical Cancer; Adaptive Radiotherapy
Keywords: Cervical Cancer; Moderated Hypofractionated Radiotherapy; Adaptive Radiotherapy; Randomized controlled trial
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Experimental group (Experimental): Radiotherapy +Concurrent Chemotherapy or Immunotherapy Experimental
  Interventions: Combination Product: Moderated hypofractionated online adaptive radiotherapy
- Control group (Active Comparator): Radiotherapy +Concurrent Chemotherapy or Immunotherapy Standard of Care
  Interventions: Combination Product: Conventional radiotherapy

INTERVENTIONS:
Combination Product: Moderated hypofractionated online adaptive radiotherapy — Radiation: Moderated hypofractionated online adaptive radiotherapy (oART)+ High-dose rate (HDR) Brachytherapy
  Experimental group: 43.35Gy/17F external beam radiotherapy with oART + HDR-Brachytherapy
  Drug: Concurrent Chemotherapy or immunotherapy
  Weekly cisplatin 40 mg/m2 or PD-1 inhibitors
  Arms: Experimental group
Combination Product: Conventional radiotherapy — Radiation: External beam radiotherapy (EBRT) + High-dose rate (HDR) Brachytherapy
  Contral group: 45Gy/25F EBRT + HDR-Brachytherapy
  Drug: Concurrent Chemotherapy or immunotherapy
  Weekly cisplatin 40 mg/m2 or PD-1 inhibitors
  Arms: Control group

SUMMARY:
The most common external beam radiotherapy fractionation scheme for cervical cancer is 45-50.4 Gy delivered in 25-28 fractions. However, prolonged treatment duration can lead to insufficient availability of medical resources. We hope to assess the safety and efficacy of moderated hypofractionated online adaptive radiotherapy in combination with brachytherapy in patients with cervical cancer in a multicenter study.

DETAILED DESCRIPTION:
This is a multicenter, non-inferiority, phase 3, randomized controlled study. This study investigates the role of moderated hypofractionated online adaptive radiotherapy by randomizing patients to this experimental regimen versus the standard of treatment.The purpose of this study is to access safety and efficacy of moderated hypofractionated online adaptive radiotherapy in combination with high-dose-rate brachytherapy in patients with cervical cancer, which based on the previous research (NCT05994300).

ELIGIBILITY:
Inclusion Criteria:

1. The patient is fully voluntary and has the capacity for autonomy, signing the informed consent form 30 days prior to enrollment
2. Age ≥18 and ≤75 years
3. FIGO stage IB-IIIB cervical cancer; IIIC1 (lymph node metastasis ≤2 cm, without common iliac lymph node metastasis)
4. Pathologically diagnosed as squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma
5. Concurrent weekly cisplatin therapy ± immunotherapy
6. Able to undergo brachytherapy
7. ECOG performance status of 0-1, with an expected ability to tolerate lying flat for half an hour.

Exclusion Criteria:

1. Patients who have undergone cervical cancer surgery, excluding pelvic lymphadenectomy or pelvic lymph node dissection, or cervical conization
2. FIGO stages IA, IIIC2, IVA, or IVB
3. FIGO stage IIIC1 with lymph nodes >2 cm, or with common iliac lymph node metastasis
4. History of prior abdominal or pelvic radiotherapy
5. Pregnant or breastfeeding women
6. Patients with active infections or fever
7. Other severe diseases that may significantly affect clinical trial compliance, such as unstable heart disease, kidney disease, chronic hepatitis requiring treatment, poorly controlled diabetes, or mental disorders.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 3 years
  Defined as time from date of randomization to date of progression, date of death from any cause, or date of last follow-up, whichever occurs first. Cancer progression can be identified during physical exam, biopsy, or imaging of any kind.

SECONDARY OUTCOMES:
Acute toxicity | 3 months
  This outcome is assessed by physicians during each follow-up appointment, and scored according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 . Clinically relevant toxicities of gastrointestinal, genitourinary, vaginal and non-specific general symptoms (i.e. fatigue, malaise and pain) will be collected. Hematological disorders will also be collected through weekly blood work checks. Acute toxicities will be collected at baseline, and then weekly during radiotherapy/chemoradiotherapy and at 3 months after completion of radiation.
Late toxicity | 3 years
  Late toxicities will be collected from 3 months after completion of radiation onwards until the end of follow-up.
Overall survival | 3 years
  Defined as time from date of randomization to date of death from any cause, or date of last follow-up, whichever occurs first.
Quality of life (QoL) | 3 years
  QoL will evaluated by the EORTC QLQ-C30 questionnaire.QLQ-C30 questionnaire is used for all cancers and has several symptom scales, five functional scales (physical, emotional, social, role, cognitive) and a global health status scale. Response options are a four-point Likert scale from "not at all" to "very much" or a seven-point Likert scale from "very poor" to "excellent."
Quality of Life (QoL) | 3 years
  QoL will be measured by the cervical cancer module (QLQ-CX24). QLQ-CX24 includes cancer - and treatment - related items and symptoms regarding sexuality. Acute and late vaginal and sexual QoL will be assessed using the QLQ-CX24 vaginal and sexual domains respectively.
  The QLQ-CX24 responses are regarding function and symptoms of sexual and vagina health. It is based on a scale of 1 (not at all) to 4 (very much).
Locoregional progression-free survival | 3 years
  Defined as time from date of randomization to date of locoregional progression, date of death from any cause, or date of last follow-up, whichever occurs first.
Tumor response evaluation Complete remission rate | 3 months
  Evaluated with RECIST 1.1
Metastasis-free survival | 3 years
  Defined as time from date of randomization to date of development of metastasis, date of death from any cause, or date of last follow-up, whichever occurs first.
Cervical cancer-specific survival | 3 years
  Defined as time from date of randomization to date of death attributed to cervical cancer, or date of last-follow-up, whichever occurs first.
Treatment expense | 3 months
  The treatment-related costs incurred during the course of treatment.

OTHER OUTCOMES:
Assessment of tumor regression throughout EBRT | 3 months
  To be assessed through volumetric comparison of tumor volume in the pre-EBRT and post-EBRT MRI scans.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

REFERENCES:
- [Derived] Zeng Z, Chen Y, Qiu J, Yang B, Wang Z, Meng X, Sun Y, Yan J, Hu K, Zhang F. Moderately hypofractionated online adaptive radiotherapy (SWIFT-1) in cervical cancer patients: study protocol for a multi-centered, open-label, two-arm, phase III, randomized controlled study. Radiat Oncol. 2025 Jul 16;20(1):112. doi: 10.1186/s13014-025-02688-7. PMID 40671096